## STATISTICAL ANALYSIS PLAN

Title: Multimodal Biomarker Predictors of Relapse in Major Depressive Disorder: A Hybrid

Retrospective-Prospective Cohort Study

NCT Number: Not yet available

**Document Date:** 01.12.2025

#### **Statistical Analysis Plan**

### **Analysis Block 1: MDD Biomarkers (Baseline)**

**Groups:** Recurrent vs. Non-recurrent vs. Healthy

- ANOVA or Kruskal–Wallis
- Post-hoc: Tukey/Bonferroni
- Genotype: Chi-square
  Goal: Identify baseline biomarker differences distinguishing recurrent MDD phenotype.

### **Analysis Block 2: Longitudinal Change (Prospective Group)**

Model:

Biomarker Group (Relapse/No Relapse) × Time (T0 vs T2) + Random Intercept (Subject) Using Repeated Measures ANOVA or Linear Mixed Models.

## **Expected pattern:**

- Non-relapsers: abnormal at  $T0 \rightarrow$  normalized at  $T2 \rightarrow$  similar to healthy
- Relapsers: abnormal at  $T0 \rightarrow$  remain abnormal at T2

## Analysis Block 3: Early Predictors ( $T0 \rightarrow T1$ )

- ΔP300 and ΔEEG % improvement
- Logistic regression for relapse prediction
- Point-biserial correlations with relapse

#### **Analysis Block 4: Decision Algorithm Development**

#### **Normalization Index (NI):**

For each biomarker at T2:

Z-score = (Patient T2 – Healthy Mean) / Healthy SD

#### **ROC Analysis:**

- Predictor: NI
- Outcome: Relapse (Yes/No)
- AUC  $> 0.80 \rightarrow$  strong predictor
- Cut-off = optimal Youden threshold

# **Example Interpretation:**

"If P300 latency > 320 ms at medication discontinuation, relapse risk = 85%."